CLINICAL TRIAL: NCT04792541
Title: Hyaluronan in the Treatment of Residual Pockets in Periodontitis Patients: a Randomized Controlled Clinical Trial
Brief Title: Hyaluronan in the Treatment of Residual Pockets in Periodontitis Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Responsible Party: Principal Investigator, Andreas Stavropoulos, Head of the Department of Periodontology, Malmö University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HY_residual
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): saline solution
  Interventions: Other: saline solution
- test group (Experimental): HY containing gel; GUM® Afta Clear Gel, Sunstar
  Interventions: Other: HY containing gel; GUM® Afta Clear Gel, Sunstar

INTERVENTIONS:
Other: HY containing gel; GUM® Afta Clear Gel, Sunstar
  Arms: test group
Other: saline solution
  Arms: control group

SUMMARY:
Aim To evaluate the clinical and microbiological effects of a hyaluronan (HY) as adjunct to scaling and root planning of residual pockets during supportive periodontal therapy.

Material and Methods Sixty-six chronic periodontitis, that have completed the active phase of treatment and are enrolled in a supportive periodontal therapy scheme, with 4 to 8 interproximal sites with PD ≥ 5 mm < 8 mm and presence of BoP at the revaluation examination will be randomly assigned to the test (HY containing gel) or control group. Immediately after debridement of the residual pockets the test gel (GUM® Afta Clear Gel, Sunstar) will be applied into the experimental sites by the operator. Further, the participants will be instructed to apply at the experimental sites the test gel supragingivally with an interdental brush (TePe, Malmö, Sweden), once per day after tooth brushing for the first 3 months. Subgingival gel application will be repeated at the 3-month control in persistent pockets (i.e. PD ≥ 5mm + BoP). CAL, PD, BoP, and presence of plaque will be evaluated at baseline and thereafter every 3 months (i.e., after 3, 6, 9, and 12 months). Further, subgingival microbiological samples will be collected from the 4 experimental sites at baseline, 3, 6, and 12 months. Nine periodontal pathogens (Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola, Fusobacterium nucleatum, Prevotella intermedia, Parvimonas micra, Campylobacter rectus, Eikenella corrodens), total bacterial load, and amount of Candida albicans will be determined quantitatively by real-time PCR.

DETAILED DESCRIPTION:
Aim The aim of this project is to evaluate the clinical and microbiological effects of a HY as adjunct to scaling and root planning of residual pockets during supportive periodontal therapy. The primary hypothesis is that application of HY as adjunct to debridement of residual pockets in chronic periodontitis patients results in a significantly higher number of sites with reduced risk for further disease progression (i.e. attachment loss) after debridement.

Background Hyaluronan (HY) is a naturally occurring high molecular weight glycosaminoglycan present in various body fluids and tissues, and shows bacteriostatic, fungistatic, anti-inflammatory, anti-oedematous, osteoinductive, and pro-angiogenetic properties. A recently published systematic review (Bertl et al. 2015a) of controlled studies on the use of HY in non-surgical and surgical periodontal treatment showed that HY as adjunct to non-surgical and/or surgical periodontal therapy that HY has a positive, albeit moderate, effect in favour of in terms of BOP and residual PD, compared to controls. However, due to large heterogeneity of included studies, no recommendations on the mode of application or the effect size of HY as adjunct to non-surgical and surgical periodontal treatment could be made.

Material and Methods Sixty-six chronic periodontitis, that have completed the active phase of treatment and are enrolled in a supportive periodontal therapy scheme, with 4 to 8 interproximal sites with PD ≥ 5 mm < 8 mm and presence of BoP at the revaluation examination will be randomly assigned to the test (HY containing gel) or control group. Immediately after debridement of the residual pockets the test gel (GUM® Afta Clear Gel, Sunstar) will be applied into the experimental sites by the operator. Further, the participants will be instructed to apply at the experimental sites the test gel supragingivally with an interdental brush (TePe, Malmö, Sweden), once per day after tooth brushing for the first 3 months. Subgingival gel application will be repeated at the 3-month control in persistent pockets (i.e. PD ≥ 5mm + BoP). CAL, PD, BoP, and presence of plaque will be evaluated at baseline and thereafter every 3 months (i.e., after 3, 6, 9, and 12 months).

Further, subgingival microbiological samples will be collected from the 4 experimental sites at baseline, 3, 6, and 12 months. Nine periodontal pathogens (Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Treponema denticola, Fusobacterium nucleatum, Prevotella intermedia, Parvimonas micra, Campylobacter rectus, Eikenella corrodens), total bacterial load, and amount of Candida albicans will be determined quantitatively by real-time PCR.

Significance So far any possible beneficial effect of HY containing products in the treatment of residual pockets during supportive periodontal treatment has not been assessed. It seems relevant to assess whether the positive effect of HY when applied as adjunct to scaling and root planning of residual pockets during supportive periodontal therapy, may reduce the risk for further disease progression and/or the need for periodontal surgery, compared to debridement alone.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic periodontitis
* at least 10 teeth
* 4 to 8 interproximal sites with PD ≥ 5 to < 8 mm and presence of BoP at the revaluation examination
* no molar with furcation involvement (Class II or III)
* no difference in PD > 2 mm next to the experimental site

Exclusion Criteria:

* antibiotic therapy or active periodontal treatment in the previous 6 months
* long-term use of anti-inflammatory and immunosuppressive medication
* diabetes
* pregnancy or lactatio
* need for antibiotics prophylaxis
* severe occlusal dysfunction
* orthodontic treatment
* class II or III tooth mobility
* endodontic problem

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2016-12; Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
residual periodontal pockets | 12 months
  number of experimental sites showing PD < 5 mm or no PD ≥ 5 mm + BoP

REFERENCES:
- [Derived] Bertl K, Vlachou S, Pandis N, Zampelis A, Stavropoulos A. Repeated local delivery of hyaluronic acid gel as adjunctive treatment of residual pockets in periodontitis patients undergoing supportive periodontal care. A randomized controlled clinical trial. Clin Oral Investig. 2024 Feb 20;28(2):158. doi: 10.1007/s00784-024-05505-9. PMID 38376596